CLINICAL TRIAL: NCT02793297
Title: Effects of Sourdough Fermented Rye Crisp Bread on Appetite and Postprandial Metabolic Responses: A Randomized Cross-over Trial
Brief Title: Effects of Sourdough Fermented Rye Crisp Bread on Appetite and Postprandial Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Dr. Rikard Landberg, Associate Professor, Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Barilla2
Record Dates: First submitted 2016-05-29; First posted 2016-06-08 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Appetite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- refined wheat crisp bread (Experimental): refined wheat crisp bread was served as part of a complete standardized breakfast
  Interventions: Other: refined wheat crisp bread
- sourdough fermented rye crisp bread (Experimental): Sourdough fermented rye crisp bread was served as part of a complete standardized breakfast
  Interventions: Other: sourdough fermented rye crisp bread
- unfermented rye crisp bread (Experimental): Unfermented rye crisp bread was served as part of a complete standardized breakfast
  Interventions: Other: unfermented rye crisp bread

INTERVENTIONS:
Other: refined wheat crisp bread — Refined wheat crisp bread (52 g) was served as part of a regular breakfast together with margarine (15 g), cheese (20 mg), coffee/tea (150 mL), and juice (150 mL). The amount of crisp bread was adjusted so that all arms provided a similar amount of available carbohydrate (35 g).
  Arms: refined wheat crisp bread
Other: sourdough fermented rye crisp bread — Sourdough fermented rye crisp bread (59.4 g) was served as part of a regular breakfast together with margarine (15 g), cheese (20 mg), coffee/tea (150 mL), and juice (150 mL). The amount of crisp bread was adjusted so that all arms provided a similar amount of available carbohydrate (35 g).
  Arms: sourdough fermented rye crisp bread
Other: unfermented rye crisp bread — Unfermented rye crisp bread (59.8 g) was served as part of a regular breakfast together with margarine (15 g), cheese (20 mg), coffee/tea (150 mL), and juice (150 mL). The amount of crisp bread was adjusted so that all arms provided a similar amount of available carbohydrate (35 g).
  Arms: unfermented rye crisp bread

SUMMARY:
The overall objective is to evaluate the impact of sourdough fermented crisp bread on effects on appetite and postprandial glucose and insulin responses. Beneficial effects on appetite and postprandial insulin responses have been observed, particularly for unfermented rye crisp breads in a previous study. In the present study, the investigators evaluated how the intake of sourdough fermented rye crisp breads vs. unfermented rye crisp bread as well as a control refined wheat crisp bread product may affect self-rated appetite and postprandial insulin and glucose responses in healthy men and women in a meal-study. The investigators characterized intervention products with regards to microstructural and chemical features in order to elucidate underlying mechanisms for potential effects observed on appetite and postprandial metabolic responses.

DETAILED DESCRIPTION:
Two commercial whole grain rye crisp breads processed differently (unfermented and sourdough fermented) and a refined wheat control product were tested in the study. The rye crisp bread products contained similar ingredients. All products provide similar amounts of available carbohydrates (about 30g). The total amount of test product is about 50-60g.

The specific primary aim of the study: To conduct a short-term breakfast intervention study in humans (n = 24) to compare the effect of 2 high-fiber rye crisp bread products processed in different ways (sourdough fermented or unfermented) and a refined wheat control crisp bread as part of a normal breakfast on self-rated appetite, postprandial glucose and insulin concentrations. Difference in post-prandial insulin response between products is the primary endpoint.

Secondary aim (conducted if significant effects in the primary endpoint have been demonstrated): To assess changes in hormones and their relation to self-perceived satiety, hunger and desire to eat and to differences in chemical and microstructural composition of the tested foods.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30 kg/m2
* fasting plasma glucose <6.0 mmol/L,
* fasting serum insulin <11 mE/L
* serum TSH <2.5 mIE/L
* plasma LDL <5.3 mmol/L
* fasting plasma triglycerides (p-TG) <1.8 mmol/L
* habitual consumption of breakfast, lunch and dinner

Exclusion Criteria:

* smokers
* use of medications likely to affect appetite
* medical conditions involving the gastrointestinal tract
* gluten intolerance or food allergies
* physical problems with eating
* dieting or self-reported fluctuations in body weight of more than 10% three months prior to screening recent participation in a dietary study
* pregnancy
* lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Subjective appetite assessed using an electronic visual analogue scale | 360 min after breakfast
  Participants recorded their subjective sensation of fullness and hunger using an electronic visual analogue scale

SECONDARY OUTCOMES:
Glucose | 230 minutes after breakfast
  Plasma levels
insulin | 230 minutes after breakfast
  Plasma levels
GLP-1 | 230 minutes after breakfast
  Plasma levels

IPD SHARING:
Plan to Share IPD: Undecided